CLINICAL TRIAL: NCT00335517
Title: Safety and Efficacy of DepoDur in Lumbar Spine Surgery Patients
Acronym: DepoDur
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: EKR Therapeutics, Inc (Industry)
Responsible Party: Principal Investigator, Edward Puzas, Doctor, University of Rochester
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11678
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Results first posted 2013-01-09 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Lumbar Spine Surgery
Keywords: Lumbar surgery; Surgery L3-S1; DepoDur; Post-operative pain; Pain control; Pain relief
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10mg Depodur (Experimental)
  Interventions: Drug: DepoDur
- 15mg DepoDur (Experimental)
  Interventions: Drug: DepoDur

INTERVENTIONS:
Drug: DepoDur — An epidural catheter will be placed under direct vision at the conclusion of surgery. The catheter will be advanced at least 4cm to L1 level prior to injection. Two mililiters of air will be injected through the catheter to ensure patency. Aspiration will be done to ensure no intradural injections. Then the undiluted (1 or 1.5 cc) DepoDur will be injected.

SUMMARY:
The purpose of the study is to help determine the appropriate dose of DepoDur for use in spinal surgery. The study will also assess the safety of this drug in this patient population.

DETAILED DESCRIPTION:
Patients will be recruited from the general practices of Drs. Rechtine, Rubery, Molinari, and Zeidman. An epidural catheter will be placed under direct vision at the conclusion of surgery. The catheter will be advanced at least 4 cm to L1 level prior to injection. Two milliliters of air will be injected through the catheter to ensure patency. Aspiration will then be done to ensure no intradural injections. Then the undiluted (1 or 1.5 cc) DepoDurTM will be injected.

The type of surgery will be recorded as to

1. The number of levels of surgery.
2. The number of levels fused
3. The number of levels instrumented.
4. The number of levels with an interbody fusion
5. Time to ambulate
6. Time to use oral analgesics
7. The time of DepoDur injection.
8. The amount of pain medications used in the 0-2 hour time interval after injection, 2-4 hours, and each subsequent 4 hour interval.
9. Pain scores will be recorded with vital signs. (The pain score is from 1 to 10 and is asked orally to patients. This is part of the standard of care).

In a one-to-one randomization, patients will receive either a 10 or 15 mg dose of DepoDur at the time of surgery

Each patient will be provided with a morphine PCA (patient controlled analgesia) system postoperatively and then oral analgesics as appropriate. Analgesic requirements in morphine equivalents will be recorded. Comparison between the 10 and 15 mg dose will be done as to analgesic effectiveness and safety.

Post-operative orders (for 48 hours) will include epidural narcotic protocol to include. The following post-operative orders are standard of care.

1. Patient's bedside and chart will be identified as "spinal narcotic".
2. Head of bed maintained at 30 degrees of elevation.
3. 0.4 mg of Narcan (naloxone) will be added to each liter of IV fluid
4. Counted respirations and pupil size to be included with vital signs
5. Pain scores with vital signs (The pain score is from 1 to 10 and is asked orally to patients. This is part of the standard of care).
6. Continuous pulse oxymetry measurement
7. Call House officer for respiratory rate of <8 minute or changes in saturation as measured by pulse oxymetry.

Current post-operative PCA orders usually start with 1 mg of morphine per cc with a seven to ten minute lockout. Based on work by Rawal [2-3], who demonstrated that small doses of Naloxone could help eliminate nuisance side effects of epidural narcotics such as localized pruritis, 0.4 mg of Naloxon will be added to each liter of IV fluid. Continuous pulse oxymetry should be used to monitor the patient's respiratory function for 48 hours after the last dose of the epidural narcotic. Post-operative vital signs will be obtained in the recovery room by anesthesia policy. Once the patient is transferred to the floor, vital signs would be obtained every hour for the first four hours and every four hours after that.

The standard of care involves providing patients after lumbar surgery with the best pain relief possible. This can be done in a number of different ways. The use of Duramorph has been possible for many years. It has not been used recently only because of the need to re-dose. The pain relief provided by the epidural narcotic is detailed in the literature. What will be altered through this study is the addition of the long acting epidural narcotic, DepoDur. This will potentially provide for sustained pain relief for 48 hours. Usually by 48 hours postoperatively, the patient is starting to improve to a point of being able to be maintained on oral analgesics. The remainder of the study is consistent with standard of care for epidural narcotics.

ELIGIBILITY:
Inclusion Criteria:

* All mentally competent patients over the age of 18 undergoing lumbar surgery at L3-S1 who would be expected to be hospitalized for greater than 48 hours would be eligible for this study.

Exclusion Criteria:

* Patients less than 18 years old, those not able to give consent, prisoners, patients with allergies to narcotic analgesics, and pregnant women will be excluded.

Women who are pregnant or are not practicing medically acceptable contraception (a pregnancy test is used pre-operatively as part of standard of care).

Patients who experience complications during the surgery (e.g., major hemorrhage, dural puncture) will not receive the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2006-06; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rechtine Glenn, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Injection: DepoDur Injection
Period: Overall Study
Arm/Group | Injection
Started | 100
Completed | 98 (Due to pharmacy error two patients were enolled and recieved EREM, but were not included in analysis)
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Injection
Number analyzed (Participants) | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 66
  >=65 years | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 39
Region of Enrollment [Number; unit: participants]
  United States | 98

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Enrolled and Recieving Injection
Time Frame: 0-48 hours postoperatively
Measure: Number; unit: participants
Arm/Group | Injection
Number analyzed (Participants) | 98
participants | 98

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | Injection
Serious Adverse Events (participants affected / at risk) | 0/98
Other Adverse Events (participants affected / at risk) | 5/98
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Injection (N=98)
Draning Incision (Infections and infestations) | 2 (2) — 2 participants were readmitted and returned to the OR for irrigation, debridement, and reclosure of draining incision. One patient returned post operatively on day 11 and the other on day 19. All cultures were negative for infection.
Pulmonary embolus (Cardiac disorders) | 1 (1) — Patient diagnosed with a pulmonary embolus on post-op day 1. Patient had a history of atrial fibrillation treated with warfarin. Patient was treated with IVC filters and heparin anticoagulation, restarted on warfarin and discharged home.
Coronary atery disease (Cardiac disorders) | 1 (1) — One patient with a history of coronary artery disease was discharged to rehab facility where they died five days after srugery secondary to a myocardial infarction

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No